CLINICAL TRIAL: NCT04554407
Title: A Non-Randomized, Prospective Study to Evaluate the Performance of a Sustained Vacuum System
Brief Title: Study to Evaluate the Performance of a Sustained Vacuum System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SOMAVAC Medical Solutions (Industry)
Collaborators: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DOC-201419 Rev B
Record Dates: First submitted 2020-09-06; First posted 2020-09-18 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2020-09

CONDITIONS: Seroma as Procedural Complication; Hematoma Postoperative
Keywords: Seroma Following Procedure; Healing Delayed; Dehiscence

STUDY DESIGN:
Intervention Model Description: All participants receive the SOMAVAC® 100.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): All participants receive the SOMAVAC® 100 Sustained Vacuum System
  Interventions: Device: SOMAVAC® 100 Sustained Vacuum System

INTERVENTIONS:
Device: SOMAVAC® 100 Sustained Vacuum System — The SOMAVAC® 100 is a battery operated device that delivers 100mm/Hg of continuous suction.

SUMMARY:
The purpose of this study is to evaluate the performance of the SOMAVAC® 100 Sustained Vacuum System after oncologic resections.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years or older;
* Undergoing mastectomy (uni or bilateral), axillary node resection, or inguinal node resection;
* Capable of providing informed consent.

Exclusion Criteria:

* Pregnant or lactating females;
* Patients on steroids or other immune modulators known to impact healing;
* Patients who are likely to not complete the study;
* Patients who, in the opinion of the investigator, are unlikely to comply with the protocol;
* Patients who have participated in this trial previously and who were withdrawn;
* Patients with known allergies to contacting materials (i.e. latex, metal, etc.);
* Patients who received neoadjuvant chemotherapy or radiotherapy within the last 3 weeks.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Time with drains | 1 - 6 weeks
  Determine the length of time drains were used
Surgical site related complications | 1 week - 1 year
  Evaluate the number of surgical site related complication

SECONDARY OUTCOMES:
Patient reported usability of the suction device | 1week - 1year
  Determine patient reported usability of the suction device with the system usability scale
Amount of fluid collected | 1week - 6 weeks
  Determine the total amount of fluid collected

CONTACTS AND LOCATIONS:
Overall Officials: Martin D Fleming, MD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Heath Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal A, Ayantunde AA, Cheung KL. Concepts of seroma formation and prevention in breast cancer surgery. ANZ J Surg. 2006 Dec;76(12):1088-95. doi: 10.1111/j.1445-2197.2006.03949.x. PMID 17199696
- [Background] Carruthers KH, Eisemann BS, Lamp S, Kocak E. Optimizing the closed suction surgical drainage system. Plast Surg Nurs. 2013 Jan-Mar;33(1):38-42; quiz 43-4. doi: 10.1097/PSN.0b013e31828425db. PMID 23446508
- [Background] Durai R, Ng PC. How to insert a perfect chest drain. Acta Chir Belg. 2009 Oct;109(5):652-4. doi: 10.1080/00015458.2009.11680510. PMID 19994817
- [Background] Janis JE, Khansa L, Khansa I. Strategies for Postoperative Seroma Prevention: A Systematic Review. Plast Reconstr Surg. 2016 Jul;138(1):240-252. doi: 10.1097/PRS.0000000000002245. PMID 27348657
- [Background] Kuroi K, Shimozuma K, Taguchi T, Imai H, Yamashiro H, Ohsumi S, Saito S. Evidence-based risk factors for seroma formation in breast surgery. Jpn J Clin Oncol. 2006 Apr;36(4):197-206. doi: 10.1093/jjco/hyl019. PMID 16684859
- [Background] Lamp S. Closed-suction drain systems in the plastic surgery patient. Plast Surg Nurs. 2011 Oct-Dec;31(4):188-90. doi: 10.1097/PSN.0b013e318238d847. No abstract available. PMID 22157612
- [Background] Long LC. The home healthcare nurse as a patient. Home Healthc Nurse. 2013 Jan;31(1):47. doi: 10.1097/NHH.0b013e3182778da2. PMID 23238624
- [Background] Phillips BT, Wang ED, Mirrer J, Lanier ST, Khan SU, Dagum AB, Bui DT. Current practice among plastic surgeons of antibiotic prophylaxis and closed-suction drains in breast reconstruction: experience, evidence, and implications for postoperative care. Ann Plast Surg. 2011 May;66(5):460-5. doi: 10.1097/SAP.0b013e31820c0593. PMID 21407050
- [Background] Poulose BK, Shelton J, Phillips S, Moore D, Nealon W, Penson D, Beck W, Holzman MD. Epidemiology and cost of ventral hernia repair: making the case for hernia research. Hernia. 2012 Apr;16(2):179-83. doi: 10.1007/s10029-011-0879-9. Epub 2011 Sep 9. PMID 21904861
- [Background] Whitson BA, Richardson E, Iaizzo PA, Hess DJ. Not every bulb is a rose: a functional comparison of bulb suction devices. J Surg Res. 2009 Oct;156(2):270-3. doi: 10.1016/j.jss.2009.03.096. Epub 2009 May 8. PMID 19691976